CLINICAL TRIAL: NCT04337320
Title: Maternal And Neonatal Outcome of Pregnant Patients With COVID-19
Brief Title: Maternal And Neonatal Outcome of Pregnant Patients With COVID-19 in Istanbul, Turkey: A Single-Center, Retrospective, Descriptive Study
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Seda Yilmaz Semerci (Unknown)
Responsible Party: Principal Investigator, Merve Aldikactioglu Talmac, MD, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: covid19pregnancynewborn
Record Dates: First submitted 2020-04-05; First posted 2020-04-07 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Covid19; Maternal-Fetal Relations
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: newborns from covid 19 positive mothers — Evaluation of apgar, hemogram and developmental status of babies born from covid 19 positive mothers

SUMMARY:
Evaluation of apgar, hemogram and developmental status of babies born from covid 19 positive mothers

ELIGIBILITY:
Inclusion Criteria:

* from covid 19 positive mothers
* newborn mothers had not other condition or illness

Exclusion Criteria:

* from covid 19 negative mothers
* childs

Ages: 1 Minute to 15 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Evaluation of apgar, hemogram and developmental status of babies born from covid 19 positive mothers
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of apgar status of newborns from covid 19 positive mothers | 2 months
  The Apgar score is looked after at 1 and 5 minutes after birth, if the baby's Apgar score is lower than 7, it is repeated every 5 minutes until 20 minutes. Parameters examined in Apgar score Muscle tone, Heart rate, Reflexes, Skin color, Respiration.
  In the Apgar score, the baby is evaluated and scores are collected.
  7 - 10: The baby is normal.
  4 - 6: They usually recover with respiratory support.
  0 - 3: Urgent intervention and resuscitation is needed.
  The low Apgar score in the 1st minute usually returns to normal in the 5th minute with support. Despite the intervention, the Apgar scores of 5 and less at 5 and 10 minutes are associated with an increased risk of mortality and cerebral palsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)